CLINICAL TRIAL: NCT03052439
Title: Charting a Course to a Less Restrictive Diet for IBS
Brief Title: Diet Reintroduction Study in Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Shanti Eswaran, Clinical Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00122970
Record Dates: First submitted 2017-02-09; First posted 2017-02-14 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Intervention Model Description: Food items will be blindly reintroduced, and symptoms will be measured.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants blinded to randomization of order of reintroduction; Investigators blinded to order of reintroduction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Order 1 (Active Comparator): Subjects would introduce 5 different groups of FODMAPs in a blinded fashion (random order, 1 week on, one week off) while remaining on an otherwise low FODMAP diet while monitoring their IBS symptoms.
  Interventions: Other: FODMAP
- Order 2 (Active Comparator): Subjects would introduce 5 different groups of FODMAPs in a blinded fashion (random order, 1 week on, one week off) while remaining on an otherwise low FODMAP diet while monitoring their IBS symptoms.
  Interventions: Other: FODMAP
- Order 3 (Active Comparator): Subjects would introduce 5 different groups of FODMAPs in a blinded fashion (random order, 1 week on, one week off) while remaining on an otherwise low FODMAP diet while monitoring their IBS symptoms.
  Interventions: Other: FODMAP
- Order 4 (Active Comparator): Subjects would introduce 5 different groups of FODMAPs in a blinded fashion (random order, 1 week on, one week off) while remaining on an otherwise low FODMAP diet while monitoring their IBS symptoms.
  Interventions: Other: FODMAP
- Order 5 (Active Comparator): Subjects would introduce 5 different groups of FODMAPs in a blinded fashion (random order, 1 week on, one week off) while remaining on an otherwise low FODMAP diet while monitoring their IBS symptoms.
  Interventions: Other: FODMAP

INTERVENTIONS:
Other: FODMAP — After 2 weeks on a low FODMAP diet, subject will undergo a reintroduction period. 5 different FODMAPs will be reintroduced (1 week at a time, followed by 1 week washout) in a blinded, randomized fashion.

SUMMARY:
Irritable bowel syndrome (IBS) is the most common gastrointestinal disease, affecting 12% of the US population and up to 20% of the population worldwide. This is a condition that is diagnosed based on specific symptoms of altered bowel habits and abdominal pain, as well as the exclusion of select other GI diseases. IBS not only causes constipation, diarrhea, abdominal cramping, and bloating, it also significantly affects quality of life, overall functioning, and work productivity.

The cause of IBS is likely multifactorial, which makes it a difficult disease to treat. However, patients often associate their IBS symptoms with eating a meal. Up to 90% of IBS patients restrict their diet to prevent or improve their symptoms, and patients are increasingly interested in more holistic approaches to disease management. At present, the most persuasive evidence that dietary changes can treat IBS supports a diet low in fermentable carbohydrates (the low FODMAP (fermentable oligo, di, and monosaccharides and polyols) diet). This diet, which is low in certain carbohydrates, has been shown to improve IBS symptoms (particularly abdominal pain and bloating), but can be difficult to follow and quite restrictive. In addition, this diet is not meant to be used as a maintenance diet; patients undergo an elimination phase followed by a reintroduction phase of specific carbohydrate groups as they monitor their symptoms. From the results of our proposed study, the study team hopes to arrive at a modified, less -restrictive version of the low FODMAP diet that is equally effective, and also create a standard protocol that patients can use during this reintroduction phase.

Patients with IBS will be recruited into a 13-week trial that would help determine the optimal way in which high FODMAP foods should be introduced. After consent, patients would start on a low FODMAP diet for 14 days, and if their symptoms improve, they would be invited to continue in the study. For 7 days prior to the reintroduction of individual FODMAPs, patients will ingest 1daily servings of a low FODMAP nutrition drink to validate the low FODMAP content of this dietary supplement. If patients do not experience a flare of symptoms with the supplement, they enter the reintroduction period. During this period, subjects would introduce different groups of FODMAPs in a blinded fashion while remaining on an otherwise low FODMAP diet while monitoring their IBS symptoms. At the end of the study period, subjects would be informed of the FODMAPs to which they were sensitive and would meet with a dietitian. At the completion of the study, the investigators would compile the data and determine which FODMAPs were mostly likely to exacerbate IBS symptoms, thus providing the construct for a modified low FODMAP diet, or "low FODMAP-Light." It is hoped that this modified, less restrictive version of the low FODMAP diet would be equally effective for the majority of IBS patients.

DETAILED DESCRIPTION:
Research Plan Design: Blinded FODMAP reintroduction study Duration of study: 1 year

Patient population:

Eligible IBS patients

Visit 1 (-2 weeks): After providing written informed consent, baseline and descriptive data will be obtained including age, sex, race, pertinent medical history, prior IBS treatments, vital signs, weight, use of concurrent medications and supplements, duration of symptoms, and baseline symptoms. The investigators will also collect blood, stool and urine for a series of separately funded translational studies assessing immune activation, permeability, and microbiome.

After this visit, patients will enter a two-week screening period during which severity of symptoms will be assessed. Eligible patients will rate their average daily abdominal pain/discomfort as a 4 or higher on an 11 point numerical rating scale (NRS) (0-no pain, 10-intolerable pain) and IBS subtype of constipation-predominant, diarrhea- predominant, or mixed bowel habits (by Rome IV criteria19). Patients with an indeterminate subtype will be excluded. Patients will record symptoms (Table 1) daily using a web-based survey instrument. Experience from previous diet trials suggests that approximately 50% of participants will not fulfill these inclusion criteria after the screening period, and will be termed screen failures.

Visit 2 (weeks 0-2): IBS patients who fulfill the entry criteria will be invited to participate in the remainder of the trial. Instruction from an experienced research dietitian pertaining to the low FODMAP diet will be administered to all participants in an open-label fashion for 2 weeks. Patients are to continue to record symptoms daily. Our previous work has demonstrated that abdominal pain and bloating are the most responsive symptoms to the low FODMAP diet. As such, the primary measure for this study will be improvement in abdominal pain with improvement in bloating as a key secondary endpoint. If a subject experiences a ≥30% reduction in abdominal pain during the 2-week low FODMAP intervention compared to baseline, they will be invited to participate in the blinded, FODMAP reintroduction phase (below). If this ≥30% reduction is not obtained, this period of open-label low FODMAP diet will be extended an additional 2 weeks to ascertain if their symptoms improve to qualify for continuation.

Standard dietary compliance measures used in the counseling environment are to include prospectively recorded 3-day food diaries before and after the open label period. Body weight over the course of the study will also be followed. Food diaries will be analyzed for compliance via the Nutrition Data System for Research (NDSR) computer program, measuring fructose, lactose, sucrose, pectins, sorbitol, and added sugars. Blood, stool and urine samples will be collected for translational studies (separately funded).

Week 2: If a ≥30% reduction in abdominal pain is obtained from the low FODMAP diet, subjects will be eligible to continue in the study during which they will remain on a full FODMAP elimination diet. For 7 days (week 2-3) prior to the reintroduction of individual FODMAPs, subjects will ingest 1 daily servings of a low FODMAP nutrition drink (Pronourish, 170 calories each, Nestlé S.A., Vevey, Switzerland) to validate the low FODMAP content of this dietary supplement. Daily symptoms will be measured as above. If a participant does not experience a flare of symptoms with the supplement, they will continue onto the reintroduction phase. If the participant does experience a flare in symptoms, they will discontinue the product for 1 week before continuing in to the next phase (reintroduction phase) of the study. The supplement will be supplied with an unbranded label. Adverse events will be monitored during weeks 2-3 and significant adverse events (discontinuation of the supplement, worsening of GI symptoms back to baseline) will be recorded.

Visit 3 (weeks 3-13): FODMAP reintroduction (lactose, fructose, fructans, polyols, galactans) will be achieved by providing subjects with similar appearing and similar tasting snacks which will contain specific types of supplemental FODMAPs prepared by research dieticians at MCRU. The study team will ask the participants to continue on their low FODMAP diet during this reintroduction phase, with the addition of 1-2 supplemental low FODMAP drinks per day for convenience. The re-introduction of FODMAP containing foods will be conducted in a double-blind fashion where both subjects and investigators will be unaware of the type of FODMAP being reintroduced. The study dietitians will remain un-blinded to the subjects' FODMAP treatment since they will be responsible for preparing and providing the FODMAP containing supplement to the subjects. For the first 7 days of the re-introduction phase, subjects will receive a FODMAP containing food item; this treatment will be followed by a 7-day wash out period during which subjects will receive a similar food or supplement that does not contain the targeted FODMAP. The daily dose of fermentable carbohydrate contained in the study food or supplement will be administered in 2 doses (moderate for the first 3 days and higher amount for the later 4 days of the 7 day reintroduction period), with the content similar to that found in the typical American diet (internal data from healthy study subjects, published data18,20). To determine optimal dosing, the study team will conduct a careful systematic review and interviews with experienced dieticians and GIs to determine the optimal dose to each FODMAP with which to challenge. The order in which each specific FODMAP is tested will be randomized to minimize the chances of an order effect. Throughout the study period, symptom data will continue to be recorded on a daily basis (Table 1). If a subject is unable to tolerate any portion of the reintroduction phase, they will discontinue reintroduction of that specific FODMAP and revert again to a low FODMAP diet for washout.

Visit 4: Final study visit (13 weeks). Subjects will be unblinded as to which FODMAP components exacerbated symptoms, if any. This information will be disseminated to study participants by our dietitians immediately after their completion of the study period. The primary investigators remain blinded to this information through analysis of data. A three-day food diary will be obtained to ensure ongoing compliance with the low FODMAP diet. Serum samples for immune activation, stool for microbiome analysis, urine for metabolome analysis will be collected at Visit 2 and 3 and analyzed with funding from alternate sources. Body weight will again be assessed.

ELIGIBILITY:
Patient population:

Eligible non-constipated IBS (NC-IBS) patients will be invited to participate in a study that will provide double blinded, individual FODMAP challenges to patients who have responded to full dietary FODMAP restriction.

Inclusion Criteria:

* Males or females, at least 18 years of age, able to provide informed consent
* Meet Rome IV criteria for IBS-C (constipation-predominant), IBS-D (diarrhea-predominant), IBS-M (mixed bowel habits) as assessed by a gastroenterologist
* Willingness to maintain a stable dosage of IBS medications during the pretreatment baseline period, including tricyclic antidepressants; "rescue" medications permitted (ie loperamide)
* For IBS-D patients only, documentation of normal colonoscopy or flexible sigmoidoscopy with colon biopsies within five years
* Documentation of normal TSH, CBC, CRP, electrolyte panel
* Negative evaluation for celiac disease either with normal TTG IgA, EMA, and/or duodenal biopsy.

Exclusion Criteria:

* Pregnancy
* IBS-U subtype (undetermined)
* Comorbid medical problems that may affect gastrointestinal transit or motility (inflammatory bowel disease, extra-intestinal disease known to affect the gastrointestinal system (scleroderma, unstable thyroid disease, uncontrolled diabetes mellitus, etc.), severe renal or hepatic disease
* Previous treatment with a low FODMAP diet or active participation in another form of dietary therapy
* Previous surgery to the GI tract except appendectomy or cholecystectomy if performed more than six months prior to enrollment.
* Medications not permitted include probiotics, antibiotics, laxatives, and narcotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Abdominal Pain | 1 week
  Daily score (0-10) for abdominal pain will be recorded. This will be averaged and compared to the baseline and run-in periods

SECONDARY OUTCOMES:
Bloating | 1 week
  Daily score (0-10) for bloating will be recorded. This will be averaged and compared to the baseline and run-in periods
Stool Consistency | 1 week
  Daily stool consistency score will be recorded. This will be averaged and compared to the baseline and run-in periods
Stool Frequency | 1 week
  Daily number of stools will be recorded. This will be averaged and compared to the baseline and run-in periods
Stool urgency | 1 week
  Daily score (0-10) for stool urgency will be recorded. This will be averaged and compared to the baseline and run-in periods
Fatigue | 1 week
  Daily score (0-10) for fatigue will be recorded. This will be averaged and compared to the baseline and run-in periods
Sleep quality | 1 week
  Daily score (0-10) for sleep quality will be recorded. This will be averaged and compared to the baseline and run-in periods

CONTACTS AND LOCATIONS:
Overall Officials: Shanti Eswaran, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Eswaran S, Jencks KJ, Singh P, Rifkin S, Han-Markey T, Chey WD. All FODMAPs Aren't Created Equal: Results of a Randomized Reintroduction Trial in Patients With Irritable Bowel Syndrome. Clin Gastroenterol Hepatol. 2025 Feb;23(2):351-358.e5. doi: 10.1016/j.cgh.2024.03.047. Epub 2024 May 9. PMID 38729390